CLINICAL TRIAL: NCT02225275
Title: Combination of Lenalidomide and Obinutuzumab (GA101) in Patients With Recurrent Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: Lenalidomide and Obinutuzumab in Treating Patients With Recurrent or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0115; NCI-2015-00237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0115 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide, obinutuzumab) (Experimental): Patients receive obinutuzumab IV over 3-4 hours on days 1, 2, 8, and 15 of course 1 and day 1 of courses 2-6 and lenalidomide PO QD on days 9-28 of course 1 and days 1-28 of all subsequent courses. Treatment with obinutuzumab repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may continue to receive lenalidomide PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Biological: Obinutuzumab

INTERVENTIONS:
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759

SUMMARY:
This phase II trial studies how well lenalidomide and obinutuzumab work in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma that has come back (recurrent) or does not respond to treatment (refractory). Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as obinutuzumab, may interfere with the ability of cancer cells to grow and spread. Giving lenalidomide and obinutuzumab may work better in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Overall response defined as achievement of complete response (CR) or partial response (PR).

SECONDARY OBJECTIVES:

I. Safety of the combination. II. Response according to prognostic markers at diagnosis. III. Time to next treatment. IV. Overall survival.

OUTLINE:

Patients receive obinutuzumab intravenously (IV) over 3-4 hours on days 1, 2, 8, and 15 of course 1 and day 1 of courses 2-6 and lenalidomide orally (PO) once daily (QD) on days 9-28 of course 1 and days 1-28 of all subsequent courses. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may continue to receive lenalidomide PO QD in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and to provide voluntarily informed consent
* Have documented chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) according to National Cancer Institute (NCI) criteria
* Recurrent or refractory disease according to NCI criteria
* Patient are eligible if they have received one or more prior treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy > 6 months
* Serum creatinine less or equal to 2 mg/dl
* Total bilirubin less or equal to 2 mg/dl
* Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) less or equal to two times the upper normal limit
* Disease free of prior malignancies for 3 years with exception of currently treated basal cell squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast; patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in the study as long as they have a reasonable expectation to have been cured with the treatment modality received
* No prior history of myelodysplastic syndrome or other myeloid malignancy
* All participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the Revlimid REMS
* Females of childbearing potential (FCBP) must have a negative serum and/or urine pregnancy test with a sensitive of at least 50 mIU/mL within 10-14 days and again within 24 hours prior to prescribe lenalidomide for cycle 1 (prescriptions must be filled within 7 days as required by Revlimid REMS) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy

Exclusion Criteria:

* Known sensitivity to lenalidomide or other thalidomide derivatives or anti cluster of differentiation (CD)20
* Documented prolymphocytic leukemia (prolymphocytes more than 55% in the blood)
* Known history of infection with human immunodeficiency virus (HIV) or human T cell leukemia virus 1 (HTLV-1)
* Serologic status reflecting active hepatitis B or C; patients with hepatitis B (HBV) antibody positive but who have positivity for hepatitis B surface antigen (HBsAg) or anti hepatitis B core antibody (anti-HBc) and patients who are positive for anti-hepatitis C (HCV) will need to have a negative polymerase chain reaction (PCR) (viral HBV deoxyribonucleic acid [DNA] or HCV ribonucleic acid [RNA]) result prior to enrollment; those who are HBsAg positive or HBV DNA positive and those who are positive for HCV (RNA) will be excluded
* Pregnant or breast feeding females
* History of tuberculosis treated within the last five years or recent exposure to tuberculosis
* Any serious medical condition, laboratory abnormality, or psychiatric illness that places the subject unacceptable risk if he/she were to participate to the study
* Patients with a recent history of deep vein thrombosis or pulmonary embolus, in the six months prior to enrollment are not eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2016 to May 2021
Period: Overall Study
Arm/Group | Treatment (Lenalidomide, Obinutuzumab)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lenalidomide, Obinutuzumab)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 69 [60 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Response is Complete Response or Partial Response. CR is absence of Lymphadenopathy, Hepatomegaly or Splenomegaly, lymphocytes < 4000/ul, normocellular, <30% lymphocytes, no B-lymphoid nodules, Platelets > 100,000/ul, hemoglobin >11.0 g/dl and Neutrophils >1500/ul.
  PR is >/= 50% decrease in lymphadenopathy, hepatomegaly, splenomegaly and Blood Lymphocytes from baseline, 50% reduction in marrow infiltrate or B-lymphoid nodules. Platelet count > 100,000/ul, Hemoglobin > 11 g/dl and Neutrophils >1500/ul or increase >/= 50% of all over base.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide, Obinutuzumab)
Number analyzed (Participants) | 9
Participants | 5

2. Secondary Outcome: Time to Next Treatment
Description: The time-to-event outcomes (such as time to next treatment or overall survival). Time to Next Treatment is from start of study medication to the start of the next treatment, or last follow up if no next therapy.
Time Frame: Up to 5 years, 2 months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Lenalidomide, Obinutuzumab)
Number analyzed (Participants) | 9
Months | 26.9 [2.7 to 62]

3. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up. Survival will be measured by the estimated median survival computed by Kaplan-Meier (K-M) analysis, which is the time point at which the cumulative survival drops below 50%, if present. If not present then the median Overall Survival is not reached and not available (NA) as there are an insufficient number of participants with events. In either case ranges are provided for observed survival intervals used in the K-M analysis.
Time Frame: Up to 5 years, 2 months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Lenalidomide, Obinutuzumab)
Number analyzed (Participants) | 9
Months | NA [2.7 to 62] — Median not reached due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Up to 5 years, 2 months
Arm/Group | Treatment (Lenalidomide, Obinutuzumab)
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Obinutuzumab) (N=9)
Chest Pain (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fall (Injury, poisoning and procedural complications) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 2 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Obinutuzumab) (N=9)
Alanine aminiotransferase increased (Investigations) | 2 (2)
Alkaline Phosphatase Increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Aspartate Aminotransferase (Investigations) | 1 (1)
Back Pain (General disorders) | 1 (1)
Bruising (General disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Ear Inflammation (Ear and labyrinth disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 3 (4)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2)
Insomina (Psychiatric disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Lymph Node Pain (Blood and lymphatic system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Neutropenia (Investigations) | 7 (19)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (2)
Thrombocytopenia (Investigations) | 3 (7)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sclera Disorder (Eye disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT02225275/Prot_SAP_000.pdf